CLINICAL TRIAL: NCT06878014
Title: Comparison of Safety Profile and Efficacy of Different Doses of Intrathecal Morphine in Total Hip Replacement.
Brief Title: Comparing the Safety and Effectiveness of Different Doses of Morphine Administered in Spinal Anethesia for Pain Relief After Hip Replacement Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMD-01
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Analgesics, Opioid; Anesthesia, Spinal; Total Hip Replacement; Adverse Anesthesia Outcome
MeSH Terms: interventions — Anesthesia, Spinal; Bupivacaine; Acetaminophen; dexketoprofen trometamol; Dipyrone; Monitoring, Physiologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- M50 (Active Comparator): In addition to bupivacaine patients received 50 mcg morphine sulphate intrathecaly.
  Interventions: Procedure: Spinal Anesthesia (bupivacaine); Drug: Postoperative pain management with acetaminophen; Device: PCA IV Oxycodone; Drug: Postoperative pain management with dexketoprofen; Drug: Postoperative pain management with metamizole; Drug: Preemptive Analgesics; Device: Patient monitor
- M100 (Active Comparator): In addition to bupivacaine patients received 100 mcg morphine sulphate intrathecaly.
  Interventions: Procedure: Spinal Anesthesia (bupivacaine); Drug: Postoperative pain management with acetaminophen; Device: PCA IV Oxycodone; Drug: Postoperative pain management with dexketoprofen; Drug: Postoperative pain management with metamizole; Drug: Preemptive Analgesics; Device: Patient monitor
- M150 (Active Comparator): In addition to bupivacaine patients received 150 mcg morphine sulphate intrathecaly.
  Interventions: Procedure: Spinal Anesthesia (bupivacaine); Drug: Postoperative pain management with acetaminophen; Device: PCA IV Oxycodone; Drug: Postoperative pain management with dexketoprofen; Drug: Postoperative pain management with metamizole; Drug: Preemptive Analgesics; Device: Patient monitor

INTERVENTIONS:
Procedure: Spinal Anesthesia (bupivacaine) — Patients were positioned in sitting position on operating table, interspinous space was identified using anatomical landmarks (intercristal line) and palpation. Entire procedure was conducted with aseptic technique, puncture site was prepared with izopropyl alcohol solution. Skin was anesthetized with subcutaneous injection of 1% lidocaine. Spinal puncture was achieved using median or paramedian technique with 27G pencil-point spinal needle. After confirmation of free flow of cerebrospinal fluid 15 mg of 0,5% bupivacaine was administered intrathecaly. Block level was assessed by lack of sensation to alcohol swab in periumbilical area and complete motor block (Bromage 3).
Drug: Postoperative pain management with acetaminophen — Postoperatively patients received 1,0g of paracetamol every 6 hours,
Device: PCA IV Oxycodone — All patients were equipped with PCA capable syringe pump (Perfusor Space, B. Braun) with 40 milligrams of oxycodone. Care provider explained thoroughly how to operate the device and educated about possible adverse effects.
Drug: Postoperative pain management with dexketoprofen — Postoperatively patients received 50mg of dexketoprofen intravenously every 8 hours.
Drug: Postoperative pain management with metamizole — Postoperatively patients received 1,0g of metamizole intravenously every 6 hours.
Drug: Preemptive Analgesics — After securing intravenous line each patient received preemptive analgesia with 1,0g paracetamol and 1,0g metamizole.
Device: Patient monitor — Postoperatively each patient's vital signs were monitored continuously using patient monitor for 48 hours.

SUMMARY:
Pain management after total hip replacement is one of the most important aspects of postoperative care for patients and clinicians alike. One of the most common techniques used in anesthesia for this procedure is spinal anesthesia with concurrent administration of opioids into spinal sac. Addition of opioids not only prolongs the anesthesia but also provides pain relief after the procedure for a limited amount of time. Because of its unique chemical properties morphine provides the longest pain relief amongst currently known opioids lasting up to 24 hours. Unfortunately this beneficial effect is associated with both minor and serious adverse effects, most important of which is respiratory depression.

To limit this potenitialy fatal adverse effect dosing of morphine must be very precise in order to balance advantages and risks.

The aim of the study was to assess effectiveness and safety profile of different doses of morphine administered during spinal anesthesia for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in trial
* Qualification for total hip replacement surgery
* ASA physical status I-III
* BMI 19-30
* Lack of contraindications for drugs and interventions used in trial

Exclusion Criteria:

* Incapability to provide informed consent
* Contraindications for spinal anesthesia
* Preoperative chronic pain
* Chronic use of analgesics
* Obesity (BMI>30)
* Allergies and other contraindications for drugs used in trial
* Mental or physical incapability to operate PCA syringe pump

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Analgesic efficacy | 48 hours postoperatively
  Analgesic efficacy defined as mean value of NRS (Numerical Rating Scale) at 4, 8, 12 ,24 and 48 hours postoperatively at rest and during rehabilitation/movement.
Safety profile | 48 hours postoperatively
  Frequency of adverse events including excessive sedation (defined as Richmond Agitation Sedation Score RASS≤-1), constipation, postoperative nausea and vomiting, pruritus and respiratory depression defined as sudden drop in respiration rate by ≥90% for ≥10 seconds or cyanosis.

SECONDARY OUTCOMES:
Patient satisfaction | 48 hours postoperatively
  Patient satisfaction with pain management measured with Likert scale.
  1. Very satisfied.
  2. Satisfied.
  3. Neither satisfied nor dissatisfied.
  4. Dissatisfied.
  5. Very dissatisfied.
Length of stay | Up to one week.
  Length of stay postoperatively.
Time to rescue analgesia | 48 hours postoperatively
  Amount of time before first bolus of oxycodone delivered by PCA syringe pump.
Cumulative dose of oxycodone | 48 hours postoperatively
  Cumulative dose of oxycodone over 48 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Wojewódzki Szpital Specjalistyczny nr 5 im. św. Barbary, Sosnowiec, Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 1 im. prof. Tadeusza Sokołowskiego PUM w Szczecinie, Szczecin, West Pomeranian Voivodeship
  - Zespół Opieki Zdrowotnej w Końskich, Gmina Końskie, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided